CLINICAL TRIAL: NCT07224776
Title: Sparsentan for the Treatment of VEGF Signaling Pathway Inhibitor-Associated Proteinuria
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Travere Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Shruti Gupta, Director of Onconephrology, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-683
Record Dates: First submitted 2025-07-28; First posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Proteinuric Renal Disease; Proteinuric Kidney Disease; Proteinuria; Proteinuria in Nephrotic Range
Keywords: vascular endothelial growth factor inhibitors; cancer; proteinuria; endothelin-1 antagonist
MeSH Terms: conditions — Proteinuria; Neoplasms | interventions — sparsentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment with sparsentan, an endothelin-1 antagonist (Active Comparator): Participants will receive sparsentan 200 mg daily for 2 weeks, and will then titrate up to a target of 400 mg daily. After the Week 8 visit, patients will return to standard-of-care. We will compare the mean percent change in urine protein to creatinine ratio in patients treated with sparsentan versus historical controls who did not receive sparsentan.
  Interventions: Drug: sparsentan
- Historical controls with high-grade proteinuria not treated with sparsentan (Placebo Comparator): Participants must meet all eligibility criteria, but did not receive sparsentan. Historical controls will be matched based on age, sex, race, stage and cancer type
  Interventions: Drug: No sparsentan

INTERVENTIONS:
Drug: sparsentan — Participants will receive sparsentan 200 mg daily for 2 weeks, and will then titrate up to a target of 400 mg daily. Safety and feasibility will be assessed. The mean percent change in urine protein to creatinine ratio will be assessed from screening to week 8, and compared to historical controls not treated with sparsentan.
  Arms: Treatment with sparsentan, an endothelin-1 antagonist
Drug: No sparsentan — Historical controls who did not receive sparsentan, and are matched to patients who are treated with sparsentan
  Arms: Historical controls with high-grade proteinuria not treated with sparsentan

SUMMARY:
Single-center, open-label, two-stage pilot study examining the efficacy and safety of sparsentan for reducing high-grade proteinuria among patients with cancer who receive vascular endothelial growth factor inhibitors

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 18 years old) with active malignancy who are currently treated with VSPIs
2. New high-grade proteinuria, defined as ≥ 2+ proteinuria on dipstick or a calculated urinary protein-to-creatinine ratio ≥ 1.0 g/g
3. Able to provide written inform consent

Exclusion Criteria:

1. Estimated glomerular filtration rate (eGFR) < 45 ml/min/1.73m2
2. Baseline high grade proteinuria ≥ 2+ proteinuria on dipstick or a calculated urinary protein-to creatinine ratio or microalbumin-to-creatinine ≥ 1.0 g/g prior to VSPI initiation
3. Acute kidney injury defined as serum creatinine at least 1.5 times above the most proximal serum creatinine prior to VSPIs initiation
4. History of allergic reactions or angioedema to any angiotensin receptor blocker (ARB) or ERA, including sparsentan or irbesartan, or has a hypersensitivity to any of the excipients in the study medications.
5. Any potassium value >5 mEq/L in the 14 days preceding high-grade proteinuria
6. History of organ transplantation, with the exception of corneal transplants.
7. History of congestive heart failure (New York Heart Association Class II-IV)
8. History of clinically significant cerebrovascular disease (transient ischemic attack or stroke) and/or coronary artery disease (hospitalization for myocardial infarction or unstable angina, new onset of angina with positive functional tests, coronary angiogram revealing stenosis, or a coronary revascularization procedure) within 6 months prior to screening.
9. Jaundice, hepatitis, or known hepatobiliary disease (excluding asymptomatic cholelithiasis), or alanine aminotransferase and/or aspartate aminotransferase >2 times the upper limit of the normal at screening.
10. Body weight <50 kg at screening
11. Unable to hold renin-angiotensin-aldosterone system (RAAS) inhibitors such as angiotensin converting enzyme inhibitors (ACEIs), angiotensin receptor blockers (ARBs), spironolactone, eplerenone, aliskiren, aldosterone blockers during run-in period
12. Concomitant use of the following medications:

    1. Inhibitors of endothelin system such as ambrisentan, bosentan, macitentan
    2. Potassium-sparing diuretics such as amiloride, triamterene
    3. Antiarrhythmic medications such as amiodarone, digoxin
    4. Weight loss medications such as orlistat or amphetamine derivative agents
    5. St. John's wort or other hypericum-derived products
    6. Strong CYP3A inhibitors such as ketoconazole, itraconazole, posaconazole, voriconazole, clarithromycin, telithromycin, ritonavir- or cobicistat-boosted regimens, boceprevir, telaprevir, conivaptan, mibefradil
13. Pregnant or breastfeeding
14. Concurrent participation in a study with an alternative experimental therapy that may interact with sparsentan
15. Any condition that, in the view of the principal investigator, might place the patient at increased risk or compromise the integrity of the study
16. Conflict with other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in urine to protein creatinine ratio (UPCR) | 8 weeks
  The geometric mean percent change in UPCR from screening day to Week 8

SECONDARY OUTCOMES:
VSPI discontinuation or interruption | 8 weeks
  Incidence of VSPI discontinuation or interruption in the 8 weeks following onset of high-grade proteinuria
Resolution of Proteinuria | 8 weeks
  Incidence of resolution of high-grade proteinuria, defined as recovery of UPCR < 0.5 g/g in the 8 weeks following onset of high-grade proteinuria

OTHER OUTCOMES:
Incidence of treatment-related adverse events including any of the following events | 8 weeks
  1. Hyperkalemia defined as serum potassium ≥ 5.5 mmol/L on two separate occasion after ruling out measurement errors and alternative causes and despite appropriate use of diuretics and dietary modification
  2. Hypotension defined as decrease in systolic blood pressure ≥20 mm Hg or diastolic blood pressure by ≥10 mm Hg from pre-sparsentan baseline with new dizziness after excluding alternative causes unrelated to sparsentan or determined at the discretion of treating physician
  3. AKI defined as serum creatinine persistently ≥ 1.5-fold from pre-sparsentan baseline on 2 consecutive lab checks after excluding alternative causes unrelated to sparsentan or determined at the discretion of treating physician
  4. Elevated liver function test defined as newly developed AST or ALT ≥ 3 times of the ULN, with or without an elevation of total serum bilirubin ≥ 2 times ULN after sparsentan initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
This is a small, pilot study with patients with cancer receiving a specific cancer treatment.